CLINICAL TRIAL: NCT02562976
Title: OLGA Stage is More Appropriate in Predicting Early Gastric Cancer Than Endoscopic Gastric Atrophy Classification and OLGIM Stage: A Prospective Study
Brief Title: OLGA Stage is More Appropriate in Predicting Early Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Director, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjxhnk3062
Record Dates: First submitted 2015-09-22; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- early gastric cancer group: use Japanese endoscopic gastric atrophy classification, Operative Link on Gastritis Assessment (OLGA), Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM) to evaluate the severity of gastric atrophy and intestinal metaplasia in patients with early gastric cancer or high-grade neoplasia(HGN)
  Interventions: Other: gastric atrophy and intestinal metaplasia
- non-early gastric cancer group: patients diagnosed as non- gastritis, gastritis or low-grade neoplasia (LGN) by pathology were defined as non-EGC group
  Interventions: Other: gastric atrophy and intestinal metaplasia

INTERVENTIONS:
Other: gastric atrophy and intestinal metaplasia — use Japanese endoscopic gastric atrophy classification, Operative Link on Gastritis Assessment (OLGA), Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM) to evaluate the severity of gastric atrophy and intestinal metaplasia

SUMMARY:
The aim of the present study was to evaluate characteristics of background mucosa in early gastric cancer (EGC), and to seek for the optimal assessment for EGC screening.

DETAILED DESCRIPTION:
Japanese endoscopic gastric atrophy (EGA) classification, operative link on Gastritis Assessment (OLGA), operative link on intestinal metaplasia assessment (OLGIM) and gastritis pattern are used in evaluating the severity of gastritis and intestinal metaplasia in different countries, which are risk factors of gastric cancer. The aim of the present study was to evaluate characteristics of background mucosa in early gastric cancer (EGC), and to seek for the optimal assessment for EGC screening.

A prospective study was conducted encompassing EGC patients (cases) and non-EGC patients (controls). All patients were performed endoscopic examination and systematically biopsied. Outcome measures were assessed and compared, including EGA classification as well as the OLGA/OLGIM assessment. Helicobacter pylori(H. pylori) status was detected in the meantime. A stepwise logistic regression model was performed to analyze correlations between EGA, OLGA, OLGIM and EGC.

ELIGIBILITY:
Inclusion Criteria:

* The age of patients is from 40-80 years
* Must undergo esophagogastroduodenoscopy

Exclusion Criteria:

* Clinical diagnosis of advanced gastric cancer
* Post-subtotal gastrectomy
* Acute upper gastrointestinal bleeding
* Severe systemic diseases
* Lack histology

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involved consecutive patients from 40-80 years who undergoing esophagogastroduodenoscopy
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with severe gastric atrophy and/or intestinal metaplasia in early gastric cancer and non-early gastric cancer | up to 27 months
  use the Japanese endoscopic gastric atrophy (EGA) classification(it has 6 stages-C1,C2,C3,O1,O2,O3), Operative Link on Gastritis Assessment (OLGA,it has 4 stages-I,II,III,IV), and Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM,it has 4 stages-I,II,III,IV) to pick out severe gastric atrophy and/or intestinal metaplasia(EGA stage C3-O3,OLGA/OLGIM stage III-IV)

SECONDARY OUTCOMES:
correlations between Japanese endoscopic gastric atrophy (EGA) classification, Operative Link on Gastritis Assessment (OLGA), Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM) and early gastric cancer | up to 27 months
correlations between Helicobacter pylori infection and moderate-to-severe EGA classification, OLGA stage III-IV, OLGIM stage III-IV | up to 27 months
  EGA means endoscopic gastric atrophy classification,OLGA means Operative Link on Gastritis Assessment, and OLGIM means Operative Link on Gastric Intestinal Metaplasia Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Li, MD.Ph.D, Principal Investigator — Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai,China,Shanghai Institute of Digestive Disease, Shanghai